CLINICAL TRIAL: NCT02230176
Title: Antitumor Efficacy of Peptide Receptor Radionuclide Therapy With 177Lutetium -Octreotate Randomized vs Sunitinib in Unresectable Progressive Well-differentiated Neuroendocrine Pancreatic Tumor: First Randomized Phase II.
Acronym: OCCLURANDOM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-004032-30; 2013/2043 (Other: CSET number)
Record Dates: First submitted 2014-08-27; First posted 2014-09-03 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Neuroendocrine Carcinoma
MeSH Terms: conditions — Somatostatinoma | interventions — Sunitinib; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 177Lu-DOTA0-Tyr3-Octreotate or OCLU (Experimental): 7.4 GBq per injection (max: 4 injections)
  Interventions: Drug: 177Lu-DOTA0-Tyr3-Octreotate
- Sunitinib (Active Comparator): 37.5 mg/day
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib
  Arms: Sunitinib
Drug: 177Lu-DOTA0-Tyr3-Octreotate
  Arms: 177Lu-DOTA0-Tyr3-Octreotate or OCLU

SUMMARY:
This study is the first randomized, open-label, national, multicenter, phase II study assessing the efficacy and safety of OCLU in subjects with pretreated progressive pancreatic, inoperable, somatostatin receptor positive, well differentiated pancreatic neuroendocrine tumors (WDpNET). Subjects must have experienced documented progression of disease within 1 year prior to the start of the study. The control group of patients receiving Sutent will be used as internal control to assess the hypothesis of 12 months PFS equal to 35% in patients receiving Sutent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven and reviewed well differentiated malignant pancreatic sporadic NET Metastatic disease not amenable to surgical resection
* All target lesions (lesions measurable and non-measurable according to the RECIST 1.1 criteria), of a size ≥ 15 mm, twice the spatial resolution of the somatostatin receptor scintigraphy (SRS), should be positive (grade of uptake at SRS≥ 2, equal to the physiologic liver uptake) within 24 weeks prior to enrollment. Negative target lesions are acceptable if below 15mm.
* Post first line whatever the type of systemic therapy: cytotoxic chemotherapy or everolimus or somatostatine analogs… Only one line of cytotoxic chemotherapy is authorized.
* Evaluable disease according to RECIST 1.1 criteria (Appendix 2)
* Progressing disease within 12 months prior to randomization according to RECIST 1.1 criteria ;
* ECOG performance status 0-2 (appendix 9)
* Life expectancy ≥ 6 months as prognosticated by the physician
* Age ≥ 18 years, no superior limit
* Adequate bone marrow reserve (Hb > 8, neutrophils ≥ 1500/mm³ and platelets ≥80.000/mm^3)
* Effective contraception in pre-menopausal female and male patients during and for at least 6 months post-treatment.
* Patient´s signed written informed consent
* Ability to comply with the protocol procedures
* Ability to take oral medication
* Patient affiliated to a social security system or beneficiary of the same.

Exclusion Criteria:

* Large or small cell-poorly differentiated pancreatic neuroendocrine tumor according to WHO 2010 classification
* Any patient receiving treatment with short-acting Octreotide, which cannot be interrupted for 24 h before and 24 h after the administration of 177Lu-DOTA0-Tyr3-Octreotate, or any patient receiving treatment with Octreotide LAR, which cannot be interrupted for at least 6 weeks before the administration of 177Lu-DOTA0-Tyr3-Octreotate, unless OctreoScan® imaging during continued Octreotide treatment is in accordance with the inclusion criteria n°2.
* More than one line of cytotoxic chemotherapy (a patient who received the same molecules of cytotoxic chemotherapy at several times during therapeutic management is considered to have benefit from one single line of cytotoxic chemotherapy)
* Prior external beam radiation therapy to more than 25% of the bone marrow
* Urinary incontinence
* History of prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or other treated malignancies with no evidence of disease for at least five years.
* Severe renal (measured GFR according to MDRD <50ml/mn or nephrotic syndrome) or hepatic insufficiency (ALT / AST > 2.5 x ULN or ALT/AST >5 x ULN if liver function abnormalities are due to the underlying malignancy and/or total serum bilirubin > 2.5 x ULN)
* Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
* Uncontrolled diabetes mellitus as defined by a fasting blood glucose above 2 ULN
* Decompensated heart failure (ejection fraction <45%), myocardial infarction, stroke, pulmonary embolism or revascularization procedure,unstable angina pectoris, uncontrolled cardiac arrhythmia, and clinically significant bradycardia during the last 12 months.
* Hypertension that cannot be controlled despite medications (>=160/95 mmHg despite optimal medical therapy)
* Abnormal cardiac function with 12 lead ECG. Ongoing cardiac dysrhythmias of NCI CTC grade 2, atrial fibrillation of any grade, or prolongation of the QTc interval to >470 msec for males or >480 msec for females.
* Brain metastases (unless these metastases have been treated and stabilized for at least 24 weeks, prior to enrolment in the study. Patients with a history of brain metastases must have a head CTscan with contrast or MRI to document stable disease prior to enrolment in the study.)
* Pregnancy or breast feeding (see appendix 6)
* Previous treatment with the drugs under study. Prior systemic treatment with any tyrosine kinase inhibitors or anti-VEGF angiogenic inhibitors.
* Current treatment with another investigational drug.
* Treatment with potent CYP3A4 inhibitors and inducers within 7 and 12 days, respectively prior to study drug administration.
* Prior treatments with chemotherapy or immunotherapy or somatostatine analog therapy drug (except in case of functioning syndrome for somatostatine analogue therapy) or thoracic radiotherapy within 4 weeks prior to start of treatment
* Major surgery for any cause or local radiotherapy within one month prior to start of treatment
* Liver embolisation therapy within the last 3 months prior start of treatment except if progression is demonstrated and embolised lesion not used as targets
* Unrecovered toxicity from any kind of therapy
* Active or suspected acute or chronic uncontrolled disease that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration,or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-02; Primary Completion 2024-04 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
To determine the 12 months PFS | Assessed 12 months after randomization

SECONDARY OUTCOMES:
Overall Survival | Assessed every 3 months until death
Best response | Assessed every 12 weeks until progression up to 48 months
  According to RECIST V1.1

CONTACTS AND LOCATIONS:
Overall Officials: Eric BAUDIN, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France